CLINICAL TRIAL: NCT01576172
Title: A Randomized Gene Fusion Stratified Phase 2 Trial of Abiraterone With or Without ABT-888 for Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: Abiraterone Acetate and Prednisone With or Without Veliparib in Treating Patients With Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01149; NCI-2012-01149 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-2012-01919; 12-0109; CDR0000730114; UCCRC-IL057; 9012 (Other: University of Chicago Comprehensive Cancer Center); 9012 (Other: CTEP); N01CM00038 (NIH); N01CM00039 (NIH); N01CM00071 (NIH); P30CA014599 (NIH); P50CA097186 (NIH); U01CA062491 (NIH); U01CA070095 (NIH); UM1CA186691 (NIH); UM1CA186705 (NIH); UM1CA186716 (NIH)
Record Dates: First submitted 2012-04-11; First posted 2012-04-12 (Estimated); Results first posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-10

CONDITIONS: Castration-Resistant Prostate Carcinoma; Recurrent Prostate Carcinoma; Stage IV Prostate Cancer AJCC v7
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Prednisone; deltacortene; prednylidene; veliparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (abiraterone acetate and prednisone) (Active Comparator): Patients receive abiraterone acetate PO QD and prednisone PO BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Abiraterone Acetate; Other: Laboratory Biomarker Analysis; Drug: Prednisone
- Arm II (abiraterone acetate, prednisone, and veliparib) (Experimental): Patients receive veliparib PO BID on days 1-28. Patients also receive abiraterone acetate PO QD and prednisone PO BID on day 1 (day 8 of course 1). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Abiraterone Acetate; Other: Laboratory Biomarker Analysis; Drug: Prednisone; Drug: Veliparib

INTERVENTIONS:
Drug: Abiraterone Acetate — Given PO
  Other Names: CB7630; Yonsa; Zytiga
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Drug: Veliparib — Given PO
  Other Names: ABT-888; PARP-1 inhibitor ABT-888
  Arms: Arm II (abiraterone acetate, prednisone, and veliparib)

SUMMARY:
This randomized phase II trial studies abiraterone acetate and prednisone together with veliparib to see how well it works compared to abiraterone acetate and prednisone alone in treating patients with castration-resistant prostate cancer that has spread from the primary site to other places in the body. Androgens can cause the growth of prostate cancer cells. Antiandrogen drugs, such as abiraterone acetate, may lessen the amount of androgens made by the body. Veliparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving abiraterone acetate together with prednisone and veliparib may work better than abiraterone acetate and prednisone alone in treating patients with castration-resistant prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the role of v-ets erythroblastosis virus E26 oncogene (ETS) gene fusion as a predictive biomarker for response to hormone therapy (abiraterone [abiraterone acetate]) alone or hormone therapy plus poly adenosine diphosphate-ribose polymerase 1 (PARP-1) targeted therapy (ABT-888 [veliparib]) in patients with metastatic castration resistant prostate cancer.

II. To evaluate whether the addition of PARP-1 targeted therapy is superior to hormone therapy alone based on ETS gene fusion status.

SECONDARY OBJECTIVES:

I. Rate of prostate-specific antigen (PSA) declines. II. Objective response rate. III. Progression-free survival. IV. Evaluate the qualitative and quantitative toxicity of abiraterone acetate with and without ABT-888.

TERTIARY OBJECTIVES:

I. To determine the concordance in fusion status among prostate cancer samples from the primary site, biopsied metastasis, and circulating tumor cells (CTCs).

II. To assess if ETS fusion status in the CTCs, at baseline, 12 weeks, and disease progression (or when off study) is associated with response to therapy.

III. To evaluate if the number of CTCs, as well as the expression levels of androgen receptor, RAD51 recombinase (RAD51), and gamma-H2A histone family, member X (H2aX) foci in the CTCs at baseline, at 12 weeks, and at disease progression in all patients is associated with response to therapy.

IV. To determine the role of phosphatase and tensin homolog (PTEN) loss as a predictive biomarker of response to abiraterone, alone or in combination with ABT-888.

V. To determine the role of PARP1 activity as a predictive biomarker of response to abiraterone, alone or in combination with ABT-888.

VI. To perform next-generation sequencing for discovery of novel gene fusions in prostate cancers negative for ETS fusions.

VII. To perform germline single nucleotide polymorphism (SNP) analysis of genes involved in hormone synthesis, transport, binding, metabolism, and degradation for discovery of novel SNPs predictive of response to abiraterone, alone or in combination with ABT-888.

VIII. To determine if ETS fusion ribonucleic acid (RNA) levels in blood are predictive of response to abiraterone, alone or in combination with ABT-888.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive abiraterone acetate orally (PO) once daily (QD) and prednisone PO twice daily (BID) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive veliparib PO BID on days 1-28. Patients also receive abiraterone acetate PO QD and prednisone PO BID on day 1 (day 8 of course 1). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Have a histologic or cytologic diagnosis of prostate cancer
* Have progressive metastatic castration-resistant prostate cancer, on androgen-deprivation therapy, based on at least one of the following criteria:

  * PSA progression defined as 25% increase over baseline value with an increase in the absolute value of at least 2 ng/mL that is confirmed by another PSA level with a minimum of a 1-week interval with a minimum PSA of 2 ng/mL
  * Progression of bidimensionally measurable soft tissue (nodal metastasis) assessed within one month prior to registration by a computed tomography (CT) scan or magnetic resonance imaging (MRI) of the abdomen and pelvis
  * Progression of bone disease (evaluable disease) (new bone lesion[s]) by bone scan
* Agree to undergo a biopsy of at least 1 metastatic site for gene-fusion status analysis; adequate archival metastatic tissue can be used if available in lieu of a biopsy; patients will only be eligible for protocol therapy if the biopsy has tumor and the tissue is evaluable for ETS fusion status
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Have testosterone < 50 ng/dL; patients must continue primary androgen-deprivation with a luteinizing hormone-releasing hormone (LHRH) analogue if they have not undergone orchiectomy
* Patients must discontinue antiandrogen therapy for at least 4 weeks (e.g. flutamide, bicalutamide, nilutamide) prior to registration with no evidence of a falling PSA after washout; patients on steroids are eligible as long as they will be switched to prednisone
* Have no prior exposure to cytochrome 450 family 17(CYP-17) (other than ketoconazole) or PARP inhibitors for prostate cancer; patients with prior exposure to ketoconazole are eligible
* Patients with up to 2 prior chemotherapy regimens are eligible
* Obtained within 14 days prior to registration: White blood cells (WBC) >= 3,000/ul
* Obtained within 14 days prior to registration: Absolute neutrophil count (ANC) >= 1,500/ul
* Obtained within 14 days prior to registration: Platelet count >= 100,000/ul
* Obtained within 14 days prior to registration: Serum creatinine =< 1.5 x the institutional upper limits of normal or corrected creatinine clearance of >= 50 mg/ml/hr/1.73 m^2 body surface area (BSA)
* Obtained within 14 days prior to registration: Potassium >= 3.5 mmol/L
* Obtained within 14 days prior to registration: Bilirubin within the institutional limits of normal
* Obtained within 14 days prior to registration: Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 2 times upper limit of normal
* Obtained within 14 days prior to registration: Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 2 times upper limit of normal
* Measured within 28 days prior to administration of ABT-888: >= 10.0 g/dL hemoglobin (Hb) with no blood transfusion in the past 28 days
* Men must agree to use effective contraception during treatment and for at least 1 week after the last administration of therapy
* Patients must be able to take oral medication without crushing, dissolving, or chewing tablets
* Patients may have received prior radiation therapy or surgery; however, at least 21 days must have elapsed since completion of radiation therapy or surgery and patient must have recovered from all side effects at the time of registration
* Ability to understand and the willingness to sign a written informed-consent document that is approved by the local institutional review board

Exclusion Criteria:

* Patients may not be receiving any other investigational agents; any prior investigational products must be stopped at least 14 days (2-week washout) prior to registration
* Patients who have had chemotherapy, radiotherapy or oral antifungal agents (ketoconazole, itraconazole, fluconazole) within 3 weeks prior to entering the study or those who have not recovered (e.g. back to baseline or grade 1) from adverse events due to agents administered more than 3 weeks earlier

  * There is a potential drug interaction when abiraterone is concomitantly used with a cytochrome P450 family 2, subfamily D, polypeptide 6 (CYP2D6) substrate narrow therapeutic index (e.g., thioridazine, dextromethorphan), or strong cytochrome P450 family 3, subfamily A, polypeptide 4 [CYP3A4] inhibitors (e.g., atazanavir, erythromycin, indinavir, itraconazole, Ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, and voriconazole) or strong inducers (e.g., carbamazepine, phenobarbital, phenytoin, rifabutin, rifampin, rifapentine); caution should be used when patients are on one of these drugs
* Patients with history of active seizures are not eligible
* Patients with a history of pituitary or adrenal dysfunction, active or symptomatic viral hepatitis, or chronic liver disease are not eligible
* Patients with known brain metastases should be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ABT-888 or abiraterone
* Patients may continue on a daily multi-vitamin, calcium and vitamin D, but all other herbal, alternative and food supplements (i.e. PC-Spes, saw palmetto, St John's wort, etc.) must be discontinued before registration; patients must not be planning to receive any concurrent cytotoxic chemotherapy, surgery, or radiation therapy during protocol treatment; hormonal-acting agents (including diethylstilbestrol/DES, aldosterone, and spironolactone) are forbidden during the trial and must be stopped prior to registration; no washout period will be required for any of these agents; patients on megestrol acetate for hot flashes are allowed to continue therapy
* Patients on stable doses of bisphosphonates or denosumab which have been started prior to registration may continue on this medication, patients who are not on bisphosphonates or denosumab are eligible as long as they initiate therapy prior to registration
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (New York Heart Association class III and IV heart failure), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements or concurrent medications that alter cardiac conduction
* Patients with a "currently active" second malignancy other than non-melanoma skin cancers are not eligible; patients are not considered to have a "currently active" malignancy if they have completed all therapy and are now considered without evidence of disease for 1 year
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Patients with treatment-related acute myeloid leukemia (AML) (t-AML)/myelodysplastic syndrome (MDS) or with features suggestive of AML/MDS. Prior allogeneic bone marrow transplant or double umbilical cord blood transplantation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2012-03-30 (Actual); Primary Completion 2019-10-23 (Actual); Study Completion 2020-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maha H Hussain, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (14):
- United States (14):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - City of Hope South Pasadena, South Pasadena, California
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - M D Anderson Cancer Center, Houston, Texas
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin Women's Health Center, Madison, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

REFERENCES:
- [Derived] Hussain M, Daignault-Newton S, Twardowski PW, Albany C, Stein MN, Kunju LP, Siddiqui J, Wu YM, Robinson D, Lonigro RJ, Cao X, Tomlins SA, Mehra R, Cooney KA, Montgomery B, Antonarakis ES, Shevrin DH, Corn PG, Whang YE, Smith DC, Caram MV, Knudsen KE, Stadler WM, Feng FY, Chinnaiyan AM. Targeting Androgen Receptor and DNA Repair in Metastatic Castration-Resistant Prostate Cancer: Results From NCI 9012. J Clin Oncol. 2018 Apr 1;36(10):991-999. doi: 10.1200/JCO.2017.75.7310. Epub 2017 Dec 20. PMID 29261439

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Abiraterone Acetate and Prednisone) | Arm II (Abiraterone Acetate, Prednisone, and Veliparib)
Started | 79 | 80
Completed | 74 | 79
Not Completed | 5 | 1
Not completed — Ineligible | 2 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Insurance issue | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Abiraterone Acetate and Prednisone) | Arm II (Abiraterone Acetate, Prednisone, and Veliparib) | Total
Number analyzed (Participants) | 74 | 79 | 153
Age, Continuous [Median (Full Range); unit: years] | 69 [50 to 90] | 68 [47 to 85] | 68 [47 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 74 | 79 | 153
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 9 | 3 | 12
  White | 61 | 74 | 135
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Prostate-specific Antigen (PSA) Response Rate
Description: 50% or greater decline in PSA from baseline.
Time Frame: Up to 3 years
Population: 2 patients non-evaluable in Arm I and 3 patients non-evaluable in Arm II due to receiving <2 treatment cycles
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Abiraterone Acetate and Prednisone) | Arm II (Abiraterone Acetate, Prednisone, and Veliparib)
Number analyzed (Participants) | 72 | 76
Participants | 46 | 55
Statistical Analysis 1: Comparison: Arm I (Abiraterone Acetate and Prednisone) vs Arm II (Abiraterone Acetate, Prednisone, and Veliparib); Test type: Superiority; p = 0.27, Chi-squared

2. Secondary Outcome: Rates of PSA Decline
Description: Change in PSA from baseline to 12 weeks
Time Frame: 12 weeks
Population: 3 patients in Arm 1 and 13 patients in Arm 2 had missing data.
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Arm I (Abiraterone Acetate and Prednisone) | Arm II (Abiraterone Acetate, Prednisone, and Veliparib)
Number analyzed (Participants) | 71 | 66
ng/ml | -41.1 (15.7) | -52.9 (26.5)
Statistical Analysis 1: Comparison: Arm I (Abiraterone Acetate and Prednisone) vs Arm II (Abiraterone Acetate, Prednisone, and Veliparib); Test type: Superiority; p = 0.70, t-test, 2 sided; t=-0.39 on 112.7 degrees of freedom (Satterthwaite)

3. Secondary Outcome: Objective Response Rates in Patients With Measurable Disease.
Description: Overall response per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 3 years
Population: Subset of patients with measurable disease.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Abiraterone Acetate and Prednisone) | Arm II (Abiraterone Acetate, Prednisone, and Veliparib)
Number analyzed (Participants) | 40 | 46
Participants | 18 | 24
Statistical Analysis 1: Comparison: Arm I (Abiraterone Acetate and Prednisone) vs Arm II (Abiraterone Acetate, Prednisone, and Veliparib); Test type: Superiority; p = 0.51, Chi-squared

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Time from randomization to disease progression or death.
Time Frame: Up to 42 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Abiraterone Acetate and Prednisone) | Arm II (Abiraterone Acetate, Prednisone, and Veliparib)
Number analyzed (Participants) | 72 | 76
months | 10.1 [8.2 to 13.8] | 11.0 [8.1 to 13.6]
Statistical Analysis 1: Comparison: Arm I (Abiraterone Acetate and Prednisone) vs Arm II (Abiraterone Acetate, Prednisone, and Veliparib); Test type: Superiority; p = 0.99, Log Rank

5. Secondary Outcome: Grade 4 or 5 Adverse Events
Description: Grade 4 or greater toxicity graded by the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 at least possibly related to treatment.
Time Frame: 30 days after completion of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Abiraterone Acetate and Prednisone) | Arm II (Abiraterone Acetate, Prednisone, and Veliparib)
Number analyzed (Participants) | 74 | 79
Participants | 1 | 3
Statistical Analysis 1: Comparison: Arm I (Abiraterone Acetate and Prednisone) vs Arm II (Abiraterone Acetate, Prednisone, and Veliparib); Test type: Superiority; p = 0.62, Fisher Exact

ADVERSE EVENTS:
Time Frame: 30 days after completion of study treatment (up to 42 months).
Description: Toxicity graded by the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 without regard to attribution.
Arm/Group | Arm I (Abiraterone Acetate and Prednisone) | Arm II (Abiraterone Acetate, Prednisone, and Veliparib)
All-Cause Mortality (participants affected / at risk) | 0/74 | 1/79
Serious Adverse Events (participants affected / at risk) | 15/74 | 17/79
Other Adverse Events (participants affected / at risk) | 74/74 | 79/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Abiraterone Acetate and Prednisone) (N=74) | Arm II (Abiraterone Acetate, Prednisone, and Veliparib) (N=79)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 2
Chest pain - cardiac (Cardiac disorders) | 0 | 1
Colonic obstruction (Gastrointestinal disorders) | 1 | 0
Confusion (Psychiatric disorders) | 0 | 1
Cystitis noninfective (Renal and urinary disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 1
General disorders and administration site conditions - Other, specify (General disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Heart failure (Cardiac disorders) | 2 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1
Hypertension (Vascular disorders) | 1 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1
Hypotension (Vascular disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 2
Lung infection (Infections and infestations) | 1 | 1
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 1
Pain (General disorders) | 0 | 1
Pain in extremity (Metabolism and nutrition disorders) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 1
Renal calculi (Renal and urinary disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 2
Sepsis (Infections and infestations) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Stroke (Nervous system disorders) | 0 | 1
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 2 | 1
Urostomy obstruction (Injury, poisoning and procedural complications) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 3
Wound infection (Infections and infestations) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Abiraterone Acetate and Prednisone) (N=74) | Arm II (Abiraterone Acetate, Prednisone, and Veliparib) (N=79)
Abdominal pain (Gastrointestinal disorders) | 9 | 5
Alanine aminotransferase increased (Investigations) | 14 | 7
Alkaline phosphatase increased (Investigations) | 19 | 15
Anemia (Blood and lymphatic system disorders) | 24 | 26
Anorexia (Metabolism and nutrition disorders) | 7 | 12
Anxiety (Psychiatric disorders) | 3 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 7
Aspartate aminotransferase increased (Investigations) | 17 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 23 | 16
Blood bilirubin increased (Investigations) | 8 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 14 | 10
Bruising (Injury, poisoning and procedural complications) | 6 | 14
Constipation (Gastrointestinal disorders) | 9 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 10
Creatinine increased (Investigations) | 8 | 8
Cystitis noninfective (Renal and urinary disorders) | 3 | 6
Diarrhea (Gastrointestinal disorders) | 14 | 15
Dizziness (Nervous system disorders) | 11 | 16
Dry mouth (Gastrointestinal disorders) | 1 | 5
Dysgeusia (Nervous system disorders) | 1 | 4
Dyspepsia (Gastrointestinal disorders) | 1 | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 | 12
Edema limbs (General disorders) | 19 | 8
Fall (Injury, poisoning and procedural complications) | 8 | 7
Fatigue (General disorders) | 30 | 44
Flank pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 | 2
Headache (Nervous system disorders) | 11 | 14
Hematuria (Renal and urinary disorders) | 2 | 7
Hot flashes (Vascular disorders) | 15 | 24
Hypercalcemia (Metabolism and nutrition disorders) | 6 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 16 | 23
Hyperkalemia (Metabolism and nutrition disorders) | 11 | 6
Hypernatremia (Metabolism and nutrition disorders) | 6 | 6
Hypertension (Vascular disorders) | 18 | 15
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 | 7
Hypocalcemia (Metabolism and nutrition disorders) | 7 | 7
Hypoglycemia (Metabolism and nutrition disorders) | 7 | 5
Hypokalemia (Metabolism and nutrition disorders) | 7 | 11
Hyponatremia (Metabolism and nutrition disorders) | 15 | 9
Hypophosphatemia (Metabolism and nutrition disorders) | 17 | 14
Hypotension (Vascular disorders) | 4 | 0
Insomnia (Psychiatric disorders) | 10 | 11
Lymphocyte count decreased (Investigations) | 10 | 20
Depression (Psychiatric disorders) | 5 | 5
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 8
Nausea (Gastrointestinal disorders) | 16 | 47
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 6
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 4
Non-cardiac chest pain (General disorders) | 5 | 2
Pain (General disorders) | 12 | 21
Pain in extremity (Musculoskeletal and connective tissue disorders) | 28 | 14
Paresthesia (Nervous system disorders) | 4 | 4
Pelvic pain (Reproductive system and breast disorders) | 4 | 1
Platelet count decreased (Investigations) | 12 | 9
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 5
Sinusitis (Infections and infestations) | 4 | 2
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 5 | 4
Skin infection (Infections and infestations) | 2 | 4
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 9 | 9
Urinary frequency (Renal and urinary disorders) | 9 | 16
Urinary incontinence (Renal and urinary disorders) | 5 | 8
Urinary tract infection (Infections and infestations) | 1 | 7
Vomiting (Gastrointestinal disorders) | 7 | 18
Weight gain (Investigations) | 8 | 3
Weight loss (Investigations) | 9 | 11
White blood cell decreased (Investigations) | 4 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-24): https://cdn.clinicaltrials.gov/large-docs/72/NCT01576172/Prot_SAP_001.pdf